CLINICAL TRIAL: NCT01093729
Title: A Dose Block-randomized, Double-blind, Single Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of HM11260C After Subcutaneous Administration in Healthy Male Subjects
Brief Title: A Study of HM11260C in Healthy Male Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-EXC-101
Record Dates: First submitted 2010-03-23; First posted 2010-03-26 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Exendin-4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort1 (Experimental): HM11260C 0.5mcg/kg or Placebo
  Interventions: Drug: HM11260C
- Cohort2 (Experimental): HM11260C 2mcg/kg or Placebo
  Interventions: Drug: HM11260C
- Cohort3 (Experimental): HM11260C 4mcg/kg or Placebo
  Interventions: Drug: HM11260C
- Cohort4 (Experimental): HM11260C 8mcg/kg or Placebo
  Interventions: Drug: HM11260C
- Cohort5 (Experimental): HM11260C 14mcg/kg or Placebo
  Interventions: Drug: HM11260C

INTERVENTIONS:
Drug: HM11260C — HM11260C 0.5mcg/kg or Placebo
  Arms: Cohort1
Drug: HM11260C — HM11260C 2mcg/kg or Placebo
  Arms: Cohort2
Drug: HM11260C — HM11260C 4mcg/kg or Placebo
  Arms: Cohort3
Drug: HM11260C — HM11260C 8mcg/kg or Placebo
  Arms: Cohort4
Drug: HM11260C — HM11260C 14mcg/kg or Placebo
  Arms: Cohort5

SUMMARY:
Study Design: Randomized, double-blind, placebo-controlled, escalating single-dose design. Five ascending dose cohorts are planned.

DETAILED DESCRIPTION:
Primary Objective: To assess the safety, tolerability, pharmacokinetics and pharmacodynamics of single subcutaneous dose of HM11260C in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age range 20 to 45 years
2. Weight>50 and < 90kg, Body mass index of >18 and <27 Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study

Exclusion Criteria

1. Acute disease within 1 month prior to start of study drug administration
2. Has previously disease which affect drug absorption, distribution, metabolism, excretion (e.g., inflammatory gastric disease, gastric or intestinal ulcer, hepatic disease, renal disease)
3. History or presence of clinically significant and active cardiovascular, pulmonary, renal, endocrine, hematological, gastrointestinal, central nervous system, psychiatric disorder, autoimmune disease, or malignant tumor
4. Has unsuitable clinical test results through the medical checkup, within 35 days prior to start of administration of study drug (medical history, physical examination, ECG, laboratory test)
5. Laboratory test results

   1. AST (sGOT) or ALT (sGPT) > 1.25Xupper normal limit
   2. Total bilirubin > 1.5Xupper normal limit
   3. Absolute Neutrophil Count < 1500 mm2
6. History or presence of clinically significant allergic disease (including mild allergic rhinitis and allergic dermatitis which is not necessary to medication)
7. Prior exposure to products related to Exenatide
8. Use of any prescription medication within 14 days prior to Day 1
9. Use of any medication within 7 days prior to Day 1 (over-the-counter medication, herbal products, nutrient, vitamins)
10. Subject who can't eat standard meal received by Korea University Anam Hospital
11. Donor of whole blood for transfusion within 60 days prior to start of study drug administration or donor of apheresis within 20 days or Receiver of blood transfusion within 1 month
12. Participation in another clinical study within 60 days prior to start of study drug administration
13. Taking Caffein(> 5cups/ day) or alcohol abuse (> 30g/ day) or excessive smoker(> 10 Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety | 1, 2, 3, 4, 5, 7, 9, 16, 22, 30, 36, 43, 57, 84 Day
  Investigate Safety of HM10560A: Safety data, including physical examinations, laboratory evaluation, ECGs, vital signs, adverse events, and immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Clinical, Principal Investigator — Korea